CLINICAL TRIAL: NCT03478241
Title: Postoperative Pain Intensity Associated With the Use of Different Nickel Titanium Instrumentation Systems During Single-Appointment Non-Surgical Endodontic Retreatment: A Randomized Clinical Trial
Brief Title: Postoperative Pain Intensity Associated With the Use of Different Nickel Titanium Instrumentation Systems
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Tan Firat Eyuboglu, Assistant Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 481
Record Dates: First submitted 2018-03-14; First posted 2018-03-27 (Actual); Last update posted 2018-03-27 (Actual); Status verified 2018-03

CONDITIONS: Pain, Postoperative; Endodontically Treated Teeth
Keywords: Endodontic retreatment; postoperative pain; OneShape; Revo-S; WaveOne
MeSH Terms: conditions — Pain, Postoperative; Tooth, Nonvital

STUDY DESIGN:
Intervention Model Description: after each group has been treated with their respective Ni-Ti root canal shaping system, post operative pain was assessed at 6, 12, 18, 24, 48, and 72 h; 7 days; and 1 month.
Who Masked: Participant
Masking Description: the patient did not know which shaping system was used on them
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: single file rotary motion (Active Comparator): after the previous root canal filling was removed, the shaping procedure of the root canal system was carried out using OneShape Ni-Ti system.
  Interventions: Device: Group 1: single file rotary motion
- Group 2: multiple file rotary motion (Active Comparator): after the previous root canal filling was removed, the shaping procedure of the root canal system was carried out using Revo S Ni-Ti system.
  Interventions: Device: Group 2: multiple file rotary motion
- Group 3: single file reciprocal motion (Active Comparator): after the previous root canal filling was removed, the shaping procedure of the root canal system was carried out using WaveOne Ni-Ti system.
  Interventions: Device: Group 3: single file reciprocal motion

INTERVENTIONS:
Device: Group 1: single file rotary motion — after the previous root canal filling was removed, the shaping procedure of the root canal system was carried out using OneShape Ni-Ti system. the obturation process was completed prior to coronal restoration either with direct or indirect methods
  Other Names: OneShape
  Arms: Group 1: single file rotary motion
Device: Group 2: multiple file rotary motion — after the previous root canal filling was removed, the shaping procedure of the root canal system was carried out using Revo S Ni-Ti system. the obturation process was completed prior to coronal restoration either with direct or indirect methods
  Other Names: Revo S
  Arms: Group 2: multiple file rotary motion
Device: Group 3: single file reciprocal motion — after the previous root canal filling was removed, the shaping procedure of the root canal system was carried out using WaveOne Ni-Ti system. the obturation process was completed prior to coronal restoration either with direct or indirect methods
  Other Names: WaveOne
  Arms: Group 3: single file reciprocal motion

SUMMARY:
In this study the effect of different engine-driven nickel titanium (Ni-Ti) instrumentation systems (OneShape, Revo S and WaveOne) on postoperative dental pain in patients with asymptomatic teeth after a single-appointment root canal retreatment was evaluated.

DETAILED DESCRIPTION:
The aim of this clinical study was to evaluate the effect of different engine-driven nickel titanium (Ni-Ti) instrumentation systems (OneShape, Revo S and WaveOne) on postoperative dental pain in patients with asymptomatic teeth after a single-appointment root canal retreatment. A total of a hundred thirty nine patients with asymptomatic teeth and with no contradictory medical history who were indicated for non-surgical retreatment at the Endodontic Clinic, Faculty of Dentistry, Istanbul Medipol University, between September and December 2016 were included in this study. All of the patients have been recruited from the Istanbul Medipol University Dental Clinics in Istanbul. Out of a hundred thirty nine patients, a total of ninety-nine patients who met the inclusion criteria and agreed to participate was enrolled for the study and were divided into three groups (n=33). Consent was obtained from all study participants before the treatment. After removing previous root canal filling, instrumentation was performed using One Shape, Revo-S, and WaveOne in groups 1, 2, and 3, respectively. All retreatments were performed in a single appointment by one endodontist before permanent coronal restoration. Postoperative pain intensity was assessed at 6, 12, 18, 24, 48, and 72 h; 7 days; and 1 month after the retreatment. The teeth was examined according to for pain intensity, percussion & palpation sensitivity, swelling, analgesic intake and clinical status.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic teeth
* Patients with no contradictory medical history
* Patients who were indicated for non-surgical retreatment and
* Patients who were above 18 years old

Exclusion Criteria:

* Patients aged below 18 years;
* Symptomatic teeth,
* Teeth with vertical root fractures
* Teeth with excessive periodontal disease;
* Patients who received or required surgical endodontic treatment
* Patients diagnosed with systemic diseases
* Patients who used analgesics 12 h before or
* Patients who used antibiotics 1 month before the retreatment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Postoperative Pain after single appointment retreatment at 1 month | 6, 12, 18, 24, 48, and 72 h; 7 days; and 1 month
  The primary outcome measure of the study was to assess if different nickel titanium root canal shaping systems influence the intensity and duration of postoperative pain in single-visit non-surgical root canal re-treatments. Postoperative pain was recorded using a four-level verbal rating scale, where 0 indicated no pain, 1 indicated slight pain, 2 indicated moderate pain, and 3 indicated sever pain. the patients were asked to return to the clinic for assessing postoperative pain (tenderness to palpation and percussion) at 24, 48, and 72 h; 7 days; and 1 month after the treatment. One clinician performed all the assessments at 24, 48, and 72 h; 7 days; and 1 month.

OTHER OUTCOMES:
unscheduled appointment for emergency intervention | 1 month
  the presence or absence of unscheduled appointment for emergency dental intervention was recorded on the chart of the patient as "present" or "absent" during the observation time
presence of complications | 1 month
  the absence or presence of complications (such as swelling or parasthesia) after the intervention was recorded on the chart of the patient as "present" or "absent" during the observation time

CONTACTS AND LOCATIONS:
Overall Officials: TAN FIRAT EYUBOGLU, DDS, PhD, Principal Investigator — Medipol University

IPD SHARING:
Plan to Share IPD: No